CLINICAL TRIAL: NCT01030679
Title: To Investigate the Glycemic Control and Lipid Profile of CKD-501 Monotherapy in Patients With Type 2 Diabetes Mellitus:a Eight-week, Multicenter, Randomized, Double-blind, Parallel-Group, Placebo-controlled, Dose-ranging Study.
Brief Title: Evaluate the Glycemic Control of CKD-501 in Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Chin Kim/Medical Director, Chong Kun Dang
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19DM05L
Record Dates: First submitted 2009-12-09; First posted 2009-12-11 (Estimated); Last update posted 2009-12-16 (Estimated); Status verified 2009-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, type 2; Glitazone
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — lobeglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- CKD-501 0.5mg (Experimental)
  Interventions: Drug: CKD-501 0.5mg
- CKD-501 1mg (Experimental)
  Interventions: Drug: CKD-501 1mg
- CKD-501 2mg (Experimental)
  Interventions: Drug: CKD-501 2mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CKD-501 0.5mg — 0.5 mg/tablet, orally, 1 tablet once daily for 8 weeks
  Other Names: Lobeglitazone
  Arms: CKD-501 0.5mg
Drug: CKD-501 1mg — 1 mg/tablet, orally, 1 tablet once daily for 8 weeks
  Other Names: Lobeglitazone
  Arms: CKD-501 1mg
Drug: CKD-501 2mg — 2 mg/tablet, orally, 1 tablet once daily for 8 weeks
  Other Names: Lobeglitazone
  Arms: CKD-501 2mg
Drug: Placebo — orally, 1 tablet once daily for 8 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of three doses of CKD-501 compared to placebo in lowering fasting plasma glucose levels in people with type 2 diabetes for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Type Ⅱ diabetes mellitus
* Fasting Plasma Glucose(FPG)≥ 126 and ≤ 270
* HbA1c between 7 and 11%
* Body mass index (BMI) in the range 21-40
* The patients who has been taking oral hypoglycemic agent or diet therapy before minimum 1 month
* Agreement with written informed consent

Exclusion Criteria:

* Type I diabetes, gestational diabetes or secondary diabetes
* Treatment with insulin(over 1month) within 3 months
* Fasting Plasma Glucose level is over 270 mg/dl
* Triglyceride level is 500 mg/dl and over
* Uncontrollable hypertension
* History of myocardial infarction, heart failure, cerebral infarction, hematencephalon or unstable angina within 6 months
* Severe hepatic dysfunction: AST, ALT, Total bilirubin, ALP level over or equal to 3 times as high as upper normal limit(UNL)
* Severe renal dysfunction: Renal failure or serum creatinine greater than 30% normal limit
* Needs treatment for acute disease, uncontrolled other diseae or diabetic complications
* In treatment concomitant drug having severe risk drug interaction with investigational drug
* History of cancer within 5 years
* History of drug abuse or alcoholism
* Hepatitis B Antigen(HBsAg) test is positive
* Treatment systemic or inhalant corticosteroids within 1 month prior to Screening
* Patient who have experience such as hypersensitivity reaction, serious adverse event or no effect by treatment with glitazones
* Fertile women who not practice contraception with appropriate methods Pregnant women or nursing mothers
* Has a contraindication to treatment investigational drug from the medical and psychogenic side
* Participated in other trial within 4 weeks Participating in other trial at present
* An impossible one who participates in clinical trial by legal or investigator's decision

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2007-07; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in fasting plasma glucose at 8 weeks | 8 weeks

SECONDARY OUTCOMES:
Change from baseline in Glycemic parameters after 8 weeks | 8 weeks
Change from baseline in Lipid parameters after 8 weeks | 8 weeks
Adverse event profile after 8 weeks of treatment | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dongseop Choi, MD.,Ph.D., Study Chair — The Korea University Anam Hospital
Locations (8):
- South Korea (8):
  - The Inje University Medical Center, Busan
  - The Yeungnam University Hospital, Daegu
  - The Chtholic University of Korea Uijeongbu St. Mary's Hospital, Gyeonggi-do
  - The Seoul National Univertisy Bundang Hospital, Gyeonggi-do
  - The Wonju Christian Hospital, Kangwon-Do
  - The Inje University Sanggye-Paik Hospital, Seoul
  - The Korea University Anam Hospital, Seoul
  - The Samsung Medical Center, Seoul